CLINICAL TRIAL: NCT00726791
Title: Efficacy of rTMS (Repetitive Transcranial Magnetic Stimulation) on Patients With Somatoform Pain Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: patient did not enroll
Sponsor: Samsung Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Bum-Hee Yu, M.D. Ph.D. / Professor, Department of Psychiatry, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2008-02-071
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Pain
Keywords: chronic pain; pain disorder
MeSH Terms: conditions — Pain; Chronic Pain; Somatoform Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): high frequency rTMS applied to the motor cortex
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — Patients receive high frequency rTMS applied to the motor cortex (M1 area). The treatment protocol consists of 10 sessions of rTMS. At each session, patients receive 30 stimulation trains (10 Hz, 4 sec, 100% motor threshold) with 26 sec inter-train interval, resulting in a total of 1200 pulses per session.

SUMMARY:
Chronic somatoform pain is common in psychiatric patients. Chronic somatoform pain causes significant distress and disrupts social functioning. Moreover, chronic somatoform pain often does not sufficiently respond to medication.

Chronic somatoform pain is associated with medial pain system. The medial pain system is comprised of structures engaged in affect and motivation, such as medial thalamus and limbic structures. The medial pain system gets inhibitory control from motor cortex. Functional neuroimaging studies indicate that chronic somatoform pain is associated with hypoactivity of motor cortex, defective inhibitory process, and hyperactivity of medial pain system.

Repetitive Transcranial Magnetic Stimulation (rTMS) is a safe and non-invasive tool to modulate neurophysiologic activity of the focal brain. Therefore, pain relief by rTMS can be obtained from motor cortex stimulation, restoration of defective inhibitory process, and deactivation of medial pain system. Studies have shown that motor cortex stimulation using rTMS can relieve pain in patients with neuropathic pain. However, to our knowledge, there is no rTMS study on chronic somatoform pain in psychiatric patients. The purpose of this study is to evaluate the effect of motor cortex rTMS on chronic somatoform pain.

DETAILED DESCRIPTION:
Chronic somatoform pain is common in psychiatric patients. Chronic somatoform pain causes significant distress and disrupts social functioning. Moreover, chronic somatoform pain often does not sufficiently respond to medication.

Chronic somatoform pain is associated with medial pain system. The medial pain system is comprised of structures engaged in affect and motivation, such as medial thalamus and limbic structures. The medial pain system gets inhibitory control from motor cortex. Functional neuroimaging studies indicate that chronic somatoform pain is associated with hypoactivity of motor cortex, defective inhibitory process, and hyperactivity of medial pain system.

Repetitive Transcranial Magnetic Stimulation (rTMS) is a safe and non-invasive tool to modulate neurophysiologic activity of the focal brain. Therefore, pain relief by rTMS can be obtained from motor cortex stimulation, restoration of defective inhibitory process, and deactivation of medial pain system. Studies have shown that motor cortex stimulation using rTMS can relieve pain in patients with neuropathic pain. However, to our knowledge, there is no rTMS study on chronic somatoform pain in psychiatric patients. The purpose of this study is to evaluate the effect of motor cortex rTMS on chronic somatoform pain.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of somatoform pain disorder, chronic

Exclusion Criteria:

* Neurological disorder
* history of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The short form McGill Pain Questionnaire | baseline, mid-TMS, and after-TMS

SECONDARY OUTCOMES:
functional brain MRI | baseline and after-TMS
Clinical Global Impression | baseline, mid-TMS, and after-TMS
Hamilton Depression and Anxiety Rating Scales | baseline, mid-TMS, and after-TMS

CONTACTS AND LOCATIONS:
Overall Officials: Bum-Hee Yu, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea